CLINICAL TRIAL: NCT06552741
Title: Screening, Evaluation, and Assessment (SEA) Protocol at the NIDA IRP
Brief Title: Screening, Evaluation and Assessment (SEA) Protocol at the NIDA IRP
Status: Recruiting | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001868; 001868-DA
Record Dates: First submitted 2024-08-07; First posted 2024-08-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01-12

CONDITIONS: Substance Use Disorder; Alcohol Use Disorder
Keywords: Alcohol; Drug; Smoking; Substance; Opioid; Nicotine; Cocaine; CONTROL; Vaping
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Smoking; Vaping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Subjects without substance use disorders
- Patient: Patient with substance use disorders

SUMMARY:
Background:

People who will participate in research studies need to undergo proper screening, evaluation, and assessment (SEA). SEA helps keep those who participate in studies safe. It also helps ensure accurate study results. The National Institute on Drug Abuse (NIDA) Intramural Research Program (IRP) wants to screen people with alcohol and/or substance use disorders (ASUD) as well as people without ASUD for ongoing studies at NIDA in Baltimore, MD

Objective:

To screen people with or without ASUD for ongoing studies at NIDA. The ultimate goals are to learn why some people (1) use drugs; (2) stop using drugs; (3) use drugs but do not get addicted; and (4) never use drugs snd to develop ASUD treatments.

Eligibility:

People aged 18 years and older. They may (1) currently use nicotine, alcohol, opioids, cocaine, or other drugs; (2) no longer use them; or (3) have never used them.

Design:

Participants will have 1 screening visit that could last up to 8 hours. The visit may be split over more than 1 day. The duration of the screening may vary for each individual based on which studies they are interested in and screened for. The tests they undergo may vary and may include the following:

* Physical exam.
* Blood, saliva, and urine tests.
* Breath samples that test for alcohol and carbon monoxide.
* Test of heart function.
* Smell test that measures sense of smell.
* Tests of memory, attention, and thinking.
* Mental health evaluation.
* Mock magnetic resonance imaging (MRI) scan.
* Questionnaires about alcohol and other drug use, mental health, medical history, and life in general.

DETAILED DESCRIPTION:
Study Description:

This protocol describes the screening and evaluation process used by the National Institute on Drug Abuse (NIDA) Intramural Research Program (IRP) to assess eligibility of individuals interested in enrolling in other NIDA IRP clinical research protocols. This protocol and clinical research protocols conducted at the NIDA IRP seek to improve understanding about of the nature of alcohol and Substance Use Disorders (hereby referenced as SUD, inclusive of alcohol use disorder), determine the potential use of novel SUD therapies and establish the effects of SUD on the development, maturation, function, and structure of the body s organ systems.

Objectives:

Primary Objective:

-To provide an initial clinical and general evaluation of participants to assess eligibility for potential inclusion into other clinical research protocols at the NIDA IRP.

Secondary Objectives:

* To use the data collected for the Primary Objective toward the development and execution of hypotheses-driven and hypotheses-generating analyses.
* To create a registry of participants that may be interested in and eligible to enroll/re-enroll in NIDA IRP clinical research protocols.

Endpoints:

Primary Endpoint:

-Screening, evaluation, and assessment for eligibility to participate in other NIDA clinical research protocols.

Secondary Endpoints:

-Use the data collected for the primary endpoint to conduct future research to further characterize and understand alcohol and drug use, addiction, abstinence, and other outcomes in people with and without SUD

ELIGIBILITY:
* INCLUSION CRITERIA:

This protocol is seeking individuals with current or past SUDs and/or AUD, as well as those who have never had an SUD or AUD. These individuals also may or may not be in treatment for their AUD/SUDs.

To be eligible to participate in this study, an individual must meet the following criteria:

* Age 18-99 years old.
* Proficient ability to read, write, and understand English.
* Stated willingness to comply with all screening procedures and availability for the duration of the screening period
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Individuals who lack capacity to consent to research participation to this protocol as determined by the Evaluation to Sign Consent (ESC).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10,000 people with and without substance use disorders (SUDs), aged 18-99
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2045-01-01 (Estimated); Study Completion 2047-01-01 (Estimated)

PRIMARY OUTCOMES:
To provide an initial clinical and general evaluation of participants to assess eligibility for potential inclusion into other clinical research protocols at the NIDA IRP. | One or more visits
  To screen participants for clinical research protocols and reduce variability as well as the burden of providing the same samples and data more than once (i.e., in screening and then again in the research protocol); Eligibility for clinical research protocols can only be determined once screening requirements for a clinical research protocol(s) are completed.

SECONDARY OUTCOMES:
To use data collected for the Primary Objective to develop and execute hypotheses-driven and hypotheses-generating analyses. To create a registry of participants that may be interested in and eligible to enroll/re-enroll in NIDA clinical ... | Use the data collected for the primary endpoint to conduct future research to further characterize and understand alcohol and drug use, addiction, abstinence, and other outcomes in people with and without SUD.
  To generate data that may be used in future analyses (to be reviewed and approved as appropriate prior to commencing) in order to again maximize the utility of data and specimens while minimizing risk to subjects since no new procedures will need to be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Leggio, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choi S, Rosenbloom D, Stein MD, Raifman J, Clark JA. Differential Gateways, Facilitators, and Barriers to Substance Use Disorder Treatment for Pregnant Women and Mothers: A Scoping Systematic Review. J Addict Med. 2022 May-Jun 01;16(3):e185-e196. doi: 10.1097/ADM.0000000000000909. PMID 34380985
- [Background] Bilgin R, Tukel SS. Effects of glucose on the activity of erythrocyte membrane Ca2+ATPase in subjects with normal and impaired glucose tolerance. Biochem Mol Biol Int. 1996 Jun;39(3):547-52. doi: 10.1080/15216549600201601. PMID 8828806
- [Background] Robinson SM, Sobell LC, Sobell MB, Leo GI. Reliability of the Timeline Followback for cocaine, cannabis, and cigarette use. Psychol Addict Behav. 2014 Mar;28(1):154-62. doi: 10.1037/a0030992. Epub 2012 Dec 31. PMID 23276315
- [Background] Sobell LC, Brown J, Leo GI, Sobell MB. The reliability of the Alcohol Timeline Followback when administered by telephone and by computer. Drug Alcohol Depend. 1996 Sep;42(1):49-54. doi: 10.1016/0376-8716(96)01263-x. PMID 8889403
- [Background] Vinson DC, Reidinger C, Wilcosky T. Factors affecting the validity of a Timeline Follow-Back interview. J Stud Alcohol. 2003 Sep;64(5):733-40. doi: 10.15288/jsa.2003.64.733. PMID 14572197
- [Background] Wesson DR, Ling W. The Clinical Opiate Withdrawal Scale (COWS). J Psychoactive Drugs. 2003 Apr-Jun;35(2):253-9. doi: 10.1080/02791072.2003.10400007. PMID 12924748
- [Background] Gossop M. The development of a Short Opiate Withdrawal Scale (SOWS). Addict Behav. 1990;15(5):487-90. doi: 10.1016/0306-4603(90)90036-w. PMID 2248123
- [Background] Bohn MJ, Babor TF, Kranzler HR. The Alcohol Use Disorders Identification Test (AUDIT): validation of a screening instrument for use in medical settings. J Stud Alcohol. 1995 Jul;56(4):423-32. doi: 10.15288/jsa.1995.56.423. PMID 7674678
- [Background] Russell J, Richardson N, Dar A. Use of a modified Clinical Institute Withdrawal Assessment (CIWA) for symptom-triggered management of alcohol withdrawal syndrome. Clin Med (Lond). 2015 Jun;15 Suppl 3:s20. doi: 10.7861/clinmedicine.15-3-s20. Epub 2015 May 29. No abstract available. PMID 26026014
- [Background] Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). Br J Addict. 1989 Nov;84(11):1353-7. doi: 10.1111/j.1360-0443.1989.tb00737.x. PMID 2597811
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Wolfensberger M, Schnieper I, Welge-Lussen A. Sniffin'Sticks: a new olfactory test battery. Acta Otolaryngol. 2000 Mar;120(2):303-6. doi: 10.1080/000164800750001134. PMID 11603794
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673